CLINICAL TRIAL: NCT02148510
Title: Oral Appliance in the Treatment of Obstructive Sleep Apnea. A Randomized Controlled Blinded Multicenter Study Comparing the Efficacy of Two Devices
Brief Title: Oral Appliance in Obstructive Sleep Apnea. A Randomized Controlled Blinded Multicenter Study Comparing Two Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Apnea-2; Ethical approval # (Registry Identifier: DNR 2014/021)
Record Dates: First submitted 2014-05-16; First posted 2014-05-28 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: human; sleep apnea; adults; oral appliance; efficacy; safety; polygraphy; bruxism; cost
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Bruxism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monobloc (Experimental): Treatment with an appliance that holds the lower jaw in a fixed protruded position
  Interventions: Device: Monobloc
- Bibloc (Active Comparator): Bibloc device where a maxillary splint is connected to a mandibular splint by a connector allowing a slight opening of the jaw without compromizing the protrusion (Narval)
  Interventions: Device: Bibloc

INTERVENTIONS:
Device: Monobloc — Construction fitted to upper and lower jaw
  Other Names: Mandibular protruding device
  Arms: Monobloc
Device: Bibloc — Biblock construction
  Other Names: Narval
  Arms: Bibloc

SUMMARY:
The hypothesis of the study is that a bibloc-apnea splint has a comparable efficacy on respiratory measures as a monobloc-apnea splint and that the cost of treatment is the same. The goal is primarily to compare the Apnea-Hypopnea Index (AHI) after 6 weeks of treatment and the cost of treatment during one year.

This randomized controlled parallel group multicenter study includes 316 subjects referred for the treatment of moderate to severe Obstructive Sleep Apnea (OSA). The subjects visit the clinic at 5 scheduled occasions.

DETAILED DESCRIPTION:
The study includes 2 arms. Secondary measures are obtained by respiratory analysis and questionnaires. Electromyography (EMG) of the masseter muscle is recorded and the influence of bruxism is evaluated in terms effect on efficacy and adverse events

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of obstructive sleep apnea with AHI > 15
* Odontological status that allows retention of oral devices and with at least one molar in each quadrant
* Maximal protrusion >6 mm
* Subject giving his/her informed concent
* Understands and can communicate in Swedish
* Subject understands the instruction on how to put on the polygraphy equipment at home
* Valid AHI data at baseline respiratory analysis

Exclusion Criteria:

* age< 18 år
* BMI >35
* Jaw complaints requiring treatment the past year
* Pain or locking of the jaw at the enrollment visit
* At the discretion of the investigator judged not being able to attach to the study directives
* Hypersensitive to the material of the devices
* Ongoing Continuous Positive Airway Pressure (CPAP) treatment or oral device treatment or such treatment terminated within a month from enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Apnoea-Hypopnea-Index (AHI) | 9 weeks after start of study
  AHI defined by American Academy of Sleep Medicine (AASM)

SECONDARY OUTCOMES:
Oxygen Desaturation Index (ODI) | 9 weeks
  Number of episodes per hour with arterial oxygen saturation decline of 3% or more
Sleepiness | 9 weeks and 1 year
  Epworth Sleepiness Scale (ESS)
Quality of life | 9 weeks and 1 year
  Functional Outcomes of Sleep Questionnaire (FOSQ )
Sleep bruxism | 9 weeks
  Bruxism episodes during sleep
Adverse events | 1 year
  Subject reported and objective investigator observed events

OTHER OUTCOMES:
Cost of care | 1 year
  Total cost calculation including the device, repairs and adjustments and consumption of dentist time

CONTACTS AND LOCATIONS:
Overall Officials: Goran Isacsson, assoc prof, Study Chair — Västmanlands County hospital Västerås, Sweden
Locations (2):
- Sweden (2):
  - Västmanland County Hospitals, Västerås, Västmanland County
  - Postgraduate Dental Education Center, Örebro

REFERENCES:
- [Derived] Isacsson G, Nohlert E, Fransson AMC, Bornefalk-Hermansson A, Wiman Eriksson E, Ortlieb E, Trepp L, Avdelius A, Sturebrand M, Fodor C, List T, Schumann M, Tegelberg A. Use of bibloc and monobloc oral appliances in obstructive sleep apnoea: a multicentre, randomized, blinded, parallel-group equivalence trial. Eur J Orthod. 2019 Jan 23;41(1):80-88. doi: 10.1093/ejo/cjy030. PMID 29771314